CLINICAL TRIAL: NCT04678258
Title: A Zero Fluoroscopy Maximum Voltage Guided Stepwise Approach Using IntellaMiFi Technology Compared to Linear Ablation of the Cavotricuspid Isthmus for Typical Atrial Flutter: the ZERO MAGIC Trial
Brief Title: Zero Fluoroscopy Voltage Guided vs. Linear CTI Ablation
Acronym: ZERO MAGIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum-Fuerth (Other)
Collaborators: Boston Scientific Corporation (Industry); University of Trieste (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zero_Magic_KHF
Record Dates: First submitted 2020-12-14; First posted 2020-12-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Catheter Ablation; Atrial Flutter Typical; Radiation Exposure
Keywords: atrial flutter typical; catheter ablation; electroanatomic mapping

STUDY DESIGN:
Intervention Model Description: 2 groups, randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients are blinded to the treatment group. During FU the physician is blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: MVG ablation (Active Comparator): Group 1 - MVG: high-resolution mapping and maximum voltage guided stepwise CTI ablation (stepwise voltage guided approach (SVG)).
  Interventions: Procedure: HR electroanatomic mapping and MVG catheter ablation
- Group 2 - control: linear ablation (Active Comparator): Group 2 - control: conventional bipolar mapping and conventional linear CTI ablation.
  Interventions: Procedure: Conventional bipolar mapping and linear catheter ablation

INTERVENTIONS:
Procedure: HR electroanatomic mapping and MVG catheter ablation — High resolution CTI mapping using the mini-electrodes at the 8 mm catheter tip followed by voltage guided ablation
  Arms: Group 1: MVG ablation
Procedure: Conventional bipolar mapping and linear catheter ablation — Bipolar mapping and conventional anatomic linear catheter ablation
  Arms: Group 2 - control: linear ablation

SUMMARY:
Catheter ablation of the cavo-tricuspid isthmus (CTI) is the curative first-line therapy for typical atrial flutter. Currently, two approaches are used in clinical practice. In contrast to the conventional linear ablation approach, the Maximum voltage-guided (MVG) strategy aims to limit ablation to high voltage areas (HVAs) representing the detectable correlate of relevant conducting bundles. Data from registries show that the MVG technique is sufficient to reach comparable clinical outcome with significantly shorter ablation duration when compared to the conventional linear strategy.

Despite growing evidence, however, data from properly powered prospective randomized trials are lacking and the linear approach still remains standard. In addition, data on radiation exposure are controversial.

As a substrate-based approach, the MVG strategy requires detailed mapping and signal analysis for identification of the individual architecture and exactly targeted energy application. However, the spatial mapping resolution of large tip catheters is limited. The use of the MicroFidelity catheter technology (IntellaMiFi) with high resolution mini-electrodes at the 8 mm catheter tip can be expected to further improve the feasibility of a voltage-guided approach. In addition, the MVG approach theoretically may encompass an increased risk for clinically inapparent reconduction. A prospective study with predefined invasive re-evaluation of persistent CTI block is needed to further evaluate this issue.

Objective of this prospective randomized study is evaluate the performance of the micro-sensor technology for zero-fluoroscopy voltage-guided ablation of typical atrial flutter (AFL) compared with a population undergoing conventional linear ablation including a predefined invasive re-evaluation of persistent CTI block in addition to clinical follow-up.

The study has been approved by the responsible ethics committee.

DETAILED DESCRIPTION:
Rationale:

Catheter ablation of the CTI represents the established curative first-line treatment for typical AFl. Although the acute and chronic efficacy is high, conventional ablation is still time consuming, requires a considerable amount of radiation as reported even in the most recent trials and treatment failure occurs.

The MVG catheter ablation of the CTI aims to limit energy delivery by selectively treating conductive bundles. Compared to the conventional linear strategy, a reduction of ablation and procedural time had been shown for the MVG technique. For several reasons, however, the current evidence is still not considered to be robust enough to suggest a general change in the ablation approach:

* Despite a reduction in ablation requirements, the additional time needed for voltage mapping often prolongs the total procedure duration.
* The spatial mapping resolution of large tip catheters, most often used for CTI-ablation is limited.
* Catheter positioning and CTI ablation is still guided by fluoroscopy with the well-known potential harm in the majority of electrophysiological centers. There are conflicting data for the MVG approach regarding radiation duration.
* The MVG approach theoretically encompasses an increased risk for clinically inapparent reconduction. A prospective study with predefined invasive re-evaluation of persistent CTI block is lacking.

Aims of the study:

MicroFidelity catheter technology was introduced to enhance the spatial resolution of large tip catheters and may facilitate zero-fluoroscopy substrate-guided ablation by high-resolution (HR) electroanatomic mapping (EAM) and precisely targeted energy application.

This study is designed to prospectively evaluate safety and efficacy of the stepwise maximum voltage mapping guided CTI ablation strategy ("MVG") using IntellaMiFi technology compared with a randomized cohort undergoing conventional linear CTI ablation (control).

Beyond procedural efficacy (main hypothesis) and safety patients outcome will be evaluated

1. by electrophysiologic diagnostic reevaluation of the ablation success after 3 months,
2. by clinical assessment and Holter-monitoring during 6 and 12-month follow-up. Furthermore, we aim to validate efficacy and safety of three-dimensional EAM- guided CTI ablation without the use of fluoroscopy as standard approach in clinical routine.

The prospective randomized analysis aims to provide fundamental data to suggest a general change in the CTI ablation approach towards a three-dimensional electroanatomical mapping guided, substrate-orientated stepwise procedure without the use of radiation as clinical standard (Zero MAGIC).

Study design and hypothesis:

Single center, prospective randomized trial, two arms ("MVG": voltage mapping guided CTI ablation versus "control" undergoing linear approach), patients blinded to the treatment.

Investigators that perform follow-up will be blinded regarding the patients group.

The study is designed to prospectively compare two different ablation strategies for the curative treatment of documented typical (CTI dependent) atrial flutter regarding efficacy and safety. Patients will be randomized either to undergo a voltage mapping guided CTI ablation or to a second group ablated using the conventional linear approach in order to investigate the following hypotheses:

Main hypothesis The zero-fluoroscopy MVG ablation approach significantly reduces CTI-ablation duration (total radiofrequency (RF) energy (RFE) application time) to bidirectional conduction block (BCB) compared with the conventional linear strategy.

Further hypotheses

* Over 90% of all procedures (MVG and conventional linear) can be safely performed without the use of radiation, cardiac implantable electronic devices (CIEDs) excluded.
* IntellaMiFi electrodes localize the higher voltage potentials with higher accuracy compared to conventional bipoles.
* There is no difference in the occurrence of complications, such as tamponade, atrio-ventricular (AV) block, charring of catheter tip and sedation side effects.
* There is no difference in the rate of persistent BCB in electrophysiologic re-evaluation after 3 months.
* There is no difference in the recurrence rate of typical atrial flutter as estimated by 6 and 12 month clinical and Holter electrocardiogram follow-up.

Patients:

The trial will include consecutive patients with documented typical (CTI dependent) atrial flutter undergoing CTI ablation according to the inclusion and exclusion criteria.

Study groups and randomization Group 1 - MVG: maximum voltage guided stepwise CTI ablation (stepwise voltage guided approach (SVG)).

This cohort will be compared to Group 2 - control: patients undergoing conventional linear CTI ablation.

Primary endpoint Cumulative ablation duration (total radiofrequency energy delivery time) in seconds that is needed to achieve sustained complete BCB (acute procedural efficacy).

Secondary endpoints see below.

Follow-up Three months after ablation a diagnostic electrophysiologic (EP) study is performed to evaluate persistence of CTI block. In the case of recurrent conduction the indication is given for re-ablation.

Six and 12 months after ablation patients are invited for a clinical investigation and a 72 hours Holter monitoring is performed.

Sample size

* Primary Endpoint: procedural efficacy - ablation duration (total radiofrequency energy delivery time)

  * Primary hypothesis: MVG ablation strategy reduces the duration of RF energy application (time to CTI block) by at least 35% compared to conventional linear approach For result analysis it is planned to use a non-parametric Wilcoxon-Mann-Whitney test since the primary endpoint is not normally distributed
  * Prospective randomized trial, PROBE design
  * Group 1: treatment with MVG ablation (stepwise approach)
  * Group 2: treatment with conventional linear ablation approach
  * Sample size estimation Based on the results from Deutsch et al., Medicine 2017
* Conventional pull back/ fluoroscopy as low as reasonable achievable (ALARA): 726±454 sec.
* MVG/minimal fluoroscopy: 473±317 sec.

Compare two means two side, parametric test:

* 76 patients (2 groups with 38 pts per group)
* power 80%, α=0.05, ratio 1:1 Due to planned use of a non-parametric test 15% are added to the sample size resulting from the parametric test estimation
* Sample size: 88 patients (44 each group) plus 20% expected dropout rate: => overall sample size 106 patients (53 patients each group)

Statistics Data will be collected in a hospital-internal Excel file. The data will be initially analyzed descriptively, including frequencies and percentages for categorical data, and mean, standard deviation, median and quartiles for continuous data.

To evaluate the primary endpoint we plan to use a non-parametric Wilcoxon-Mann-Whitney test for comparison of a population not normally distributed, due to non-normality reported in former studies. We define p < 0.05 as statistically significant.

Randomization Randomization will occur once patient has been determined eligible for the study, he/she has received the appropriate and mandatory information about the study and the informed consent form has been signed. Patients will be randomly assigned with ratio 1:1 to one of two treatment arms.

The randomization list will be generated using the Wei's Urn Design method as implemented in the R package randomizeR.

Ethical consideration The study has been approved by the responsible ethics committee. In all respects, the clinical trial will be conducted in full conformance with principles of the "Declaration of Helsinki and, Good Clinical Practice (GCP).

All responsible physicians will provide a valid GCP training. All participating patients have the medical indication for curative CTI ablation according to the current medical guidelines.

Informed consent Written informed consent is required from all subjects prior to their participation in the study.

Patients insurance The study does not evaluate the performance of a medical product. All hardware and software including the catheter and EAM system are commercially available and used strictly according to their Conformité Européenne (CE) marking and specification. There is no increased radiation exposure due to the study. Despite the very low risks potentially associated to the study, a patients insurance policy will be taken out with an insurance company.

Investigator sponsored research The ZERO MAGIC trial is conducted as an investigator sponsored research (ISR) project in cooperation with Boston Scientific. The contract between the company Boston Scientific and the Klinikum Fuerth has been reviewed and approved in detail by the department for compliance from the Klinikum Fuerth.

Data management and data security The screening and informed consent process according to the inclusion and exclusion criteria will be performed by the PI and co-investigators. All participating investigators are instructed in the study protocol and provide a valid GCP training.

All demographic and procedural data will be listed in a password-protected hospital-internal Excel database according to the modified principles of the Declaration of Helsinki and Good clinical Practice. Access to the data base is restricted to the PI and co-investigators. In the data base, a cryptographic "hash" algorithm will be used for pseudonymization of patients' identifying data such as name and birth date. The code book for re-identification is password protected and the access strictly limited to Dr. Bastian, Dr. Vitali-Serdoz as PI and first co-investigator.

Data will be kept in the database for a minimum of ten years.

ELIGIBILITY:
Inclusion Criteria:

* Typical (CTI dependent) atrial flutter documented in a standard 12 lead surface ECG
* Given class I indication for curative CTI ablation according to the current guidelines
* Over 18 years old
* Given informed consent

Exclusion Criteria:

* Any contraindication for CTI ablation
* Previous CTI ablation
* BCB as procedural endpoint not assessable
* CTI ablation conducted in association with further ablation procedures
* Patients with CIED (e.g. pacemaker, ICD)
* Tricuspid valve replacement
* Right atrial thrombus
* Pregnant or breastfeeding women
* Abuse of drugs or alcohol
* Age < 18 years
* Incompliance to the treatment, e.g. necessary anticoagulation
* Expected survival less than one year
* Inability to understand the nature and rationale of the study
* Inability to take part in the follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative ablation duration | during procedure
  Cumulative ablation duration (total radiofrequency (RF) energy delivery time) in seconds that is needed to achieve sustained complete CTI block (acute procedural efficacy)

SECONDARY OUTCOMES:
Number of RF ablation points, which are necessary to achieve CTI block | during procedure
  Total number of RF ablation points with minimal local energy-delivery of 20 seconds, which are necessary to achieve CTI block
Total amount of RF energy delivery for CTI block | during procedure
  Total amount of RF energy delivery for sustained CTI block (in kilo Joules)
Rate of procedure related adverse events | during procedure
  Safety: The rate of all procedure related adverse events will be documented and analyzed
Fluoroscopy time | during procedure
  The cumulative fluoroscopy duration (in minutes)
Fluoroscopy exposure | during procedure
  Effective dose (ED in μSv)
Number of participants with persistence of CTI block | 3 months follow-up
  Number of patients with persistent bidirectional CTI block in electrophysiologic re-evaluation after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bastian, MD, Principal Investigator — Klinikum-Fuerth
Locations (1):
- Klinikum Fuerth, Fürth, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No